CLINICAL TRIAL: NCT01571973
Title: EVALUATION OF THE EFFECTIVENESS OF PHARMACEUTICAL CARE (DÁDER PROGRAM) IN DEPRESSED OUTPATIENTS TREATED WITH PSYCHOTROPIC
Brief Title: Evaluation of Pharmaceutical Care in Depressed Outpatients
Acronym: depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Regina Noto, Ph.D., Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SPPsicobio1Lu
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2011-06

CONDITIONS: Depression
Keywords: pharmaceutical care; depression; compliance; pharmacist's intervention; Dáder
MeSH Terms: conditions — Depression; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): outpatients receiving usual care
- intervention group (Experimental): outpatients receiving pharmaceutical care or pharmacotherapeutic follow-up by 6 months
  Interventions: Procedure: pharmacotherapeutic follow-up

INTERVENTIONS:
Procedure: pharmacotherapeutic follow-up — health education adjustment of dose improve compliance replacement of medication
  Arms: intervention group

SUMMARY:
The study examines whether pharmacotherapeutic follow-up improves outcomes of treatment of depressed outpatients.

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 65 years, with diagnostic hypothesis of depression at the beginning of treatment or change in treatment unless 2 months (dosage or substance)

Exclusion Criteria:

* record of dependence on psychoactive substances, diagnosed schizophrenia,
* low education (illiterate) or cognitive impairment evident that compromise the completion of research instruments

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
depression level | six months
  evaluation depression level by Beck scale

SECONDARY OUTCOMES:
anxiety level | 6 months
  evaluation anxiety level by Beck scale.
compliance | 6 months
  evaluation antidepressive treatment compliance by Morisky scale